CLINICAL TRIAL: NCT03791645
Title: Evaluating The Efficacy Of A Mind-Body Intervention In Overcoming Opioid Addiction, In Adults Undergoing Opioid Addiction Treatment
Brief Title: Evaluating The Efficacy Of A Mind-Body Intervention In Overcoming Opioid Addiction
Acronym: SKY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018H0409
Record Dates: First submitted 2018-11-07; First posted 2019-01-02 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Opioid Use; Opioid-use Disorder; Substance Use Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: SKY program includes gentle stretches, SK breathing, and cognitive coping and stressor evaluation strategies. SK breathing, the cornerstone of SKY program contains the following breathing components 1) Three-stage Ujjayi, 2) Bhastrika and 3) Rhythmic Breathing.
  Three-Stage Ujjayi is an advanced form, with each respiratory cycle lasting approximately twenty seconds. Bhastrika, involves vigorous and faster breathing, at about 20 to 30 respiratory cycles lasting 60 seconds. Three 1-minute rounds of Bhastrika are each followed by 20 seconds of normal breathing. Rhythmic breathing are slow, medium, and fast breathing cycles in succession. Respiratory rates range from about 8-12 respiratory cycles lasting approximately 10 minutes. The participant rotates through these breathing patterns.
  Upon completion of SKY program, participants will be given a home SK practice which takes approximately 25 minutes daily. Once a week, a 60-90 minutes group follow up SKY session will be held
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SKY Intervention (Experimental): Participants in the intervention group will get to participate in the SKY program, for 5 days with each day session taking 3 hours/day. SKY program involves a) specific breathing exercises and social interaction with other participants in the program. Following completion of the program, another set of questionnaires will be administered to collect information regarding stress, mood, and opioid use. After completion of the 5 day SKY program, participants will practice SKY every day at home for 30 days. They will also need to attend 4 weekly group sessions during this period and each session is expected to last 1 hour. At the end of the 30 day period, another set of questionnaires will be administered to collect information regarding stress, mood, and opioid use.
  Interventions: Behavioral: Sky Intervention
- Usual treatment (No Intervention): Participants assigned to the control group will not have access to the SKY program but will continue with usual care. They will also complete questions after 5 days and again after 30 days.

INTERVENTIONS:
Behavioral: Sky Intervention — SKY meditation has three sequential components of breathing interspersed with normal breathing. These include a) sound breath: breathing against airway resistance with slight tightening of the laryngeal muscles, (2-3 cycles/min) followed by b) bellows breath: rapid, forced expiration(20-30 cycles/min) and c) regulated, rhythmical breathing rotating through medium to fast cycles. Each session is focused upon proper breathing techniques, social interaction, and discussion of practical wisdom for everyday life to manage the mind and emotions. SKY will be administered over a 5 day period (~3 hours/day), followed by 4 weekly follow-ups (~90 min session/week) at Signature Health clinic situated in Ashtabula, Ohio.
  Arms: SKY Intervention

SUMMARY:
This study demonstrates the feasibility, acceptability of SKY program as an adjuvant therapy for American population suffering with OUD through a pilot program in Columbus, Ohio. The aim of this study is to evaluate the SKY program as an adjuvant therapy to treat opioid addiction.

DETAILED DESCRIPTION:
This research proposal aims to test the feasibility, acceptability and efficacy of SKY (Sudarshan Kriya Yoga) program, a mind-body intervention, as an adjuvant therapy for people suffering with opioid use disorder (OUD), in Columbus, Ohio. Previous research carried out in India in 2015, has demonstrated that SKY significantly improved the quality of life among people with OUD, however, the suitability, acceptability of SKY program has not been tested among American population. SKY differs from mindfulness and other meditation processes in that, it is a more physiological, rather than cognitive process. It involves controlled breathing techniques that can be easily mastered, and do not require mental effort. The investigator's goals are to a) DEMONSTRATE the feasibility, acceptability and efficacy of SKY program as an adjuvant therapy for American population suffering with OUD. Studies will be carried out in OUD subjects at Mary Haven clinic in Columbus. The efficacy of SKY will be measured using psychometric questionnaires. Feasibility and acceptability will be measured by attendance and attrition.

ELIGIBILITY:
Inclusion Criteria:

* The proposed participants are currently residents of Mary Haven
* Are currently undergoing addiction treatment which may include medication assisted treatment as well as counseling.
* The intervention is designed for adults, therefore, only individuals 18 and above will be included in the study.

Exclusion Criteria:

* Pregnant women who are beyond their first trimester are excluded from the study as the program requires breathing techniques that are not recommended for pregnant women.
* Also, patients diagnosed with schizophrenia and bipolar disorder will also be excluded from the study, as SKY program is not suitable for people with these conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in psychological health following the Sudarshan Kriya Yoga (SKY) therapy | Before SKY intervention, 1 hour after intervention and 1 month after intervention
  Change in psychological health will be measured using psychometric test administered to subjects at Signature Health clinic in Ashtabula, Ohio. The Pychometric test will involve completion of a Basic 24 Questionnaire: It is a leading behavioral health assessment tool which consists of 24 questions that cover depression and functioning.
Change in the number of participants that complete the Sudarshan Kriya Yoga (SKY) therapy | Time 1 = initial therapy session, Time 2 = week 1 post therapy session, Time 3 = week 2 post therapy session Time 4 = week 3 post therapy session, Time 5 = week 4 post therapy session Time 6 = 30 minutes daily home practice for 30 days
  To study the acceptability of the SKY program as an adjuvant therapy for American population suffering with mental disorders + opioid addiction, the attendance and attrition of the subjects at the Signature Health clinic in Ashtabula in the SKY therapy sessions will be recorded by keeping record of those that complete each progressive therapy session.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Warren, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Social Work, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No